CLINICAL TRIAL: NCT02765048
Title: Violence Prevention for Adolescent Girls With Prior Maltreatment
Acronym: GAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Missouri Department of Social Services, Children's Division (Unknown); Children's Advocacy Services of Greater St. Louis (Unknown)
Responsible Party: Principal Investigator, Wendy Auslander, Barbara A. Bailey Professor of Social Work, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201111071; R49CE001510 (NIH)
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: PTSD; Depression; Aggression; Victimization
Keywords: Adolescent girls; Child welfare; Trauma treatment; PTSD; Depression; Social problem-solving
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GAIN Program (Experimental): Subjects randomly assigned to receive the GAIN Program intervention
  Interventions: Behavioral: GAIN Program
- Usual Care (No Intervention): Subjects randomly assigned to receive community-based services as part of their usual care

INTERVENTIONS:
Behavioral: GAIN Program — Receives GAIN, a 10-session program that incorporates cognitive behavioral therapy skills in a group format to address symptoms of trauma such as PTSD and depression related to histories of child maltreatment. GAIN includes the following elements: 1) assertive communication skills and relationship boundaries, 2) understanding the connection between feelings, thoughts, and behaviors, 3) increased personal confidence, 4) how to have healthy relationships and personal safety, and 5) how to cope with stress and anxiety.
  Arms: GAIN Program

SUMMARY:
The purpose of the study is to adapt and test an evidence-based trauma treatment program for adolescent girls with histories of child maltreatment. The study adapts the CBITS (Cognitive Behavioral Intervention for Trauma in Schools) program for delivery within community-based settings for use with girls assessed and/or served by the child welfare system. The study utilizes a randomized clinical trial that evaluates the effectiveness of the adapted program entitled GAIN (Girls Aspiring toward Independence) compared with a usual care group. Primary outcomes of the intervention are mental health symptoms such as PTSD, depression, and internalizing and externalizing behaviors. Other outcomes include aggressive behaviors, revictimization, and aggression-related beliefs, self-efficacy, and behavioral intentions.

DETAILED DESCRIPTION:
Childhood maltreatment for survivors creates a risk for the perpetuation of a cycle of violence in the form of sexual violence, intimate partner violence, and child maltreatment of the next generation of children. Consistent empirical evidence across studies confirms that abuse and neglect in childhood is associated with: dating violence, serious delinquent behaviors, engaging in risky sex and substance use, physical and sexual revictimization as adult women and maltreatment as parents. Adolescent girls in foster care with histories of childhood maltreatment are at increased risk of multiple forms of interpersonal violence, as adolescents and adults, due to the presence of a multitude of additional risk factors. Mental health problems associated with the trauma of childhood maltreatment include depression, PTSD, and behavioral disorders. These problems tend to be more elevated and prevalent in adolescent girls in foster care. Additionally, these girls often experience multiple behavioral, mental health, and drug and alcohol-related problems that are also linked to interpersonal violence, suggesting that youths in foster care have different and more urgent prevention needs than other adolescents. The magnitude of the relationship between childhood maltreatment, trauma-induced mental health problems and subsequent revictimization and perpetration is so substantial and the consequences so deleterious that researchers have emphasized the necessity of targeting early intervention and prevention resources toward children exposed to violence.

There is a clear need for intervention and prevention efforts to be directed at female survivors of child maltreatment. We are targeting our intervention/prevention efforts at girls for several empirically important reasons. Prevalence studies consistently reveal that girls are more frequent victims of childhood sexual abuse, adult sexual assault and intimate partner violence. Childhood sexual abuse in particular is more strongly correlated with the development of serious mental health and substance abuse problems than other forms of maltreatment. Girls are more vulnerable to physical and sexual re-victimization in adolescence and adulthood and re-victimization increases risks of mental health and substance abuse problems, which further increases risks for re-victimization. Research has demonstrated that girls/women are more vulnerable to the development of PTSD than boys/men even when exposed to comparable levels and types of trauma, and PTSD has been shown to increase risks for re-victimization. A growing body of literature indicates that trauma responses are mediating factors in re-victimization. Consequently, if trauma symptoms (PTSD, depression, anxiety, cognitive distortions, and maladaptive coping strategies) can be ameliorated there is greater potential to prevent revictimization.

Despite the strong empirical evidence that girls with histories of maltreatment are at greater risk than other adolescents of engaging in youth violence and interpersonal violence as adults, there are no reports of violence prevention programs tailored for female adolescents in foster care. The Task Force on Community Preventive Services of the Centers for Disease Control (CDC) has identified cognitive behavior therapy as an effective treatment to reduce psychological harm among youth exposed to traumatic events and to promote healthy relationships among youths who have experienced trauma. Trauma-focused cognitive-behavioral therapy has been adapted for children exposed to community or family violence utilizing a group format and delivered in community settings. The school-based version of the intervention is known as Cognitive-Behavioral Intervention for Trauma in School, or CBITS. The study adapts the CBITS program for use with adolescent girls assessed or served by Children's Division (GAIN) who have experienced previous maltreatment for delivery within community-based settings, and evaluates its impact in preventing re-victimization and perpetration of interpersonal violence.

The specific aims of the study were to:

1. Adapt the CBITS program for girls who have been assessed or served by the Children's Division (GAIN) that targets mental health problems as they relate to risks of revictimization and perpetration of interpersonal violence.
2. Utilizing a randomized controlled design, implement the GAIN program with 125 adolescent girls who have been assessed or served by Children's Division compared with 125 girls who receive usual care.
3. Conduct a process evaluation that will monitor treatment integrity through ratings of session content delivered, participants' attendance, program relevance and satisfaction, and tracking comparison and experimental group adolescents to reduce study attrition.
4. Conduct an outcome evaluation to compare the effectiveness of the GAIN program on primary outcomes such as trauma-related mental health problems (i.e., PTSD, depression), aggression, and revictimization and on secondary outcomes such as self-efficacy to control anger and internalizing and externalizing behavior problems.

Experimental Group Youths who were randomly assigned to the experimental group participate in an informational interview conducted by a group therapist who is a licensed clinical psychologist, social worker, or counselor with extensive experience in treating girls with history of maltreatment. A significant adult chosen by the youth who is a foster parent, congregate care worker, Children's Division worker, or relative accompanied the adolescent to the informational interview so that the youth was more comfortable. The purpose of this informational interview was to inform the youth about the purpose of the group, to secure the youth's commitment to the group, to facilitate an initial connection between the adolescent and the therapist, and to assure that the youth is appropriate for the group (based on the inclusionary and exclusionary criteria). Once eligibility was determined, the therapist administered consent and assent forms.

The experimental condition consisted of the CBITS intervention adapted for adolescent girls who have been assessed or served by the Children's Division (GAIN). CBITS is an evidence-based, 10 session program that incorporates cognitive behavioral therapy skills in a group format to address symptoms of trauma, such as PTSD, anxiety, and depression related to exposure to violence. The adapted CBITS program included the following elements: psychoeducation related to common reactions to trauma, understanding the connection between feelings, thoughts, and behaviors, relaxation skills, cognitive therapy, trauma exposure, and social problem-solving. The program met once each week and lasted a total of 10 weeks. Each session was approximately 1.5 hours long. Each session had about 6-8 participants and was led by two group facilitators who had experience helping adolescents who had experienced trauma. Additionally, each participant attended two individual sessions with the group therapist to check in on her reaction to the group and to make a plan for her goals for the group. These individual sessions were an hour in length and occurred between weeks 2 and 6 of the group sessions. Following the completion of the GAIN intervention, therapists provided written recommendations to the legal custodians of experimental group participants. This report included recommendations for future care.

Experimental participants participated in three structured interviews: a pretest interview, a posttest after the intervention (approximately 3 months later), and a follow-up interview 6 months after baseline. The face-to-face pre, post, and follow-up interviews included an evaluation of the effectiveness of the GAIN program on primary and secondary outcomes. Mental health service utilization, medication use, and type and severity of child maltreatment were also assessed for potential control variables. Each interview lasted approximately one hour. Master's and doctoral level social work students conducted these face-to-face interviews. Prior to conducting interviews, interviewers participated in an intensive training to gain a working knowledge of the research project and learn to effectively discuss the risks and benefits of participation with the subjects.

Usual Care Participants Usual care participants received any usual services that they would receive during the course of the study. So for example, they continued to receive case management services through Children's Division as well as other therapeutic services as deemed appropriate by their Children's Division case manager.

Usual care participants also participated in the three evaluation interviews: a baseline interview, a posttest approximately 3 months later, and a follow-up interview 6 months after baseline. Each interview was conducted at the participant's residence or other convenient location and lasted approximately one hour. The interviews for the usual care group were similar to those administered to the experimental group participants. They included an assessment of the study's primary and secondary outcomes. Mental health service utilization, medication use, and type and severity of child maltreatment are also assessed for potential control variables.

Qualitative Follow-up Interviews Participants who were enrolled in the project after May 20, 2013 and who had not yet completed their participation in the study were invited to participate in a fourth 60-minute semi-structured qualitative interview. The purpose of the interview was to gain a deeper understanding of participants' intentions, attitudes and behaviors related to aggression as well as their experiences and perceptions of the intervention (experimental girls only), the study, and other mental health services that they have received. The qualitative interview was administered to participants (n=24) at the most convenient location for them, including their residence, Washington University, or at our collaborating agency (Children's Advocacy Services).

Semi-structured qualitative interviews were also conducted with caregivers of GAIN participants (n=17), professional staff who referred and/or worked with GAIN participants (n=8), and therapists who led the study's intervention groups (n=5). The purpose of these interviews was to gather more information about their perceptions of the youths' participation in GAIN and in other services.

Trained project staff who had experience in qualitative interviewing conducted the face-to-face interviews, which were recorded and transcribed without any identifying information. Audio files and transcripts were maintained on computer servers with all access being password protected.

ELIGIBILITY:
RCT--

Inclusion Criteria:

* Girls ages 12-18
* prior history of maltreatment that has been formally investigated and/or assessed by Children's Division
* Youth is interested in participation and provides assent through IRB approved assent forms
* The legal custodian, parent, and Family Support Team support the youth's participation and provide consent through IRB approved consent forms

Exclusion Criteria:

* Severe learning problems (i.e. can't read and/or write or cognitively impaired)
* actively suicidal or psychotic, as determined by standard protocol of the state
* behavior that would prohibit participation in a group setting or interview

Qualitative--

Caregiver and professional staff inclusion criteria are:

* Caregivers of GAIN participants (both experimental and usual care) and professional staff who referred and/or worked with GAIN participants
* Interested and willing to participate in a one-on-one interview

Exclusion criteria for caregivers and professional staff are:

-Not interested in participating in one-on-one interviews.

Therapist inclusion criteria are:

* Led the study's intervention groups with GAIN participants
* Interested and willing to participate in one-on-one interviews.

Exclusion criteria for therapists are:

-Not interested in participating in one-on-one interviews.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-08; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Child's Posttraumatic Stress Disorder Symptom Scale | Baseline to 3 months
Child Depression Inventory | Baseline to 3 months
Aggression-Problem Behavior Frequency Scale | Baseline to 3 months
Aggression-Problem Behavior Frequency Scale: Victim Version | Baseline to 3 months
Child's Posttraumatic Stress Disorder Symptom Scale | Baseline to 6 months
Child Depression Inventory | Baseline to 6 months
Aggression-Problem Behavior Frequency Scale | Baseline to 6 months
Aggression-Problem Behavior Frequency Scale: Victim Version | Baseline to 6 months

SECONDARY OUTCOMES:
Self-efficacy to Control Anger and Resolve Conflicts Scale | Baseline to 3 months
Social Problem-Solving Inventory: Revised | Baseline to 3 months
Youth Self Report: Externalizing Behaviors | Baseline to 3 months
Youth Self Report: Internalizing Behaviors | Baseline to 3 months
Self-efficacy to Control Anger and Resolve Conflicts Scale | Baseline to 6 months
Social Problem-Solving Inventory: Revised | Baseline to 6 months
Youth Self Report: Externalizing Behaviors | Baseline to 6 months
Youth Self Report: Internalizing Behaviors | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Auslander, PhD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Comtrea, Arnold, Missouri
  - Children's Advocacy Services of Greater St. Louis, St Louis, Missouri
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auslander W, Tlapek SM, Threlfall J, Edmond T, Dunn J. Mental Health Pathways Linking Childhood Maltreatment to Interpersonal Revictimization During Adolescence for Girls in the Child Welfare System. J Interpers Violence. 2018 Apr;33(7):1169-1191. doi: 10.1177/0886260515614561. Epub 2015 Nov 29. PMID 26621036
- [Background] Auslander W, Sterzing P, Threlfall J, Gerke D, Edmond T. Childhood Abuse and Aggression in Adolescent Girls Involved in Child Welfare: The Role of Depression and Posttraumatic Stress. J Child Adolesc Trauma. 2016;9:1-10. doi: 10.1007/s40653-016-0090-3. Epub 2016 Apr 12. PMID 27152132